CLINICAL TRIAL: NCT04771143
Title: A Randomized, Participant- and Investigator-blinded, Placebo-controlled, Parallel Group Study to Assess Safety, Tolerability, and Potential Interactions of Oral AFQ056 Given Concurrently With Cocaine
Brief Title: Study to Assess Safety, Tolerability, and Interactions of Cocaine and Oral AFQ056
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: study terminated/withdrawn before FPFV (no patients enrolled)
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CAFQ056A02101
Record Dates: First submitted 2021-02-24; First posted 2021-02-25 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Cocaine Use Disorder
Keywords: safety; tolerability; interaction; cocaine; cocaine use disorder; AFQ056
MeSH Terms: interventions — mavoglurant

STUDY DESIGN:
Intervention Model Description: Participants will undergo a screening infusion session with saline and cocaine on Day -2 as part of the eligibility determination. Once deemed eligible, participants will undergo screening infusion sessions 2 and 3 on Days 1 and 2 respectively. Starting Day 3, participants will receive either AFQ056 or matching placebo twice a day from Day 3 to Day 9. The AFQ056 treatment group will be up titrated to 200 mg according to the following dosing schedule: Day 3: 50 mg twice daily; Day 4: 100 mg twice daily and Days 5-9: 200 mg twice daily. On Day 10, participants will be administered only the morning dose of AFQ056 200 mg or placebo. On Days 9 and 10, participants will have infusion session 4 and 5 respectively. The participants will be discharged from the clinic on Day 12 and return for a follow-up visit between 7 to 14 days after clinic discharge. A safety follow-up call will be conducted on Day 40.
Who Masked: Participant, Investigator
Masking Description: This is a participant- and investigator-blinded study. Site staff may be unblinded to the treatment assignment of one or more participants if deemed appropriate to aid decision-making.
  Drug product will be supplied in bulk, so an unblinded pharmacy team who is independent of the study team will be required in order to maintain the blind.
  The following unblinded roles are required for this study:
  * Unblinded field monitor(s)
  * Unblinded sample analyst(s)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AFQ056 (Experimental): Experimental study drug
  Interventions: Drug: AFQ056
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AFQ056 — oral administration
  Arms: AFQ056
Drug: Placebo — matching placebo for oral administration
  Arms: Placebo

SUMMARY:
This is a study to assess safety, tolerability and interactions of AFQ056 and cocaine in patients with cocaine use disorder.

DETAILED DESCRIPTION:
This is a randomized, participant- and investigator-blinded, placebo-controlled, parallel group study to assess safety and tolerability and to compare the effects of AFQ056 on IV cocaine's physiological and subjective effects in non-treatment seeking, cocaine-experienced participants who meet American Psychiatric Association Diagnostic and Statistical Manual (DSM-V) criteria for cocaine use disorder.

Approximately twenty participants will be randomized to 2 groups (10 in each group), receiving either AFQ056 or placebo treatment for 8 days.

Participants will be screened for eligibility as outpatients and inpatients. Outpatient screening will occur between Day -28 and Day -4. On Study Day -3, participants will undergo clinic intake to screen for continued eligibility. On Study Day -2, participants will be screened for eligibility with a participant-blinded screening infusion (Infusion Session 1) of 20 mg cocaine, followed by a saline infusion, followed by a 40 mg cocaine infusion. Each 2 ml infusion of cocaine and saline will be administered by IV over a 60 second time period and approximately 60 minutes apart. Physiological and subjective data (VAS) from these sessions will be part of the eligibility criteria to continue in the study.

Once a participant has been determined to be eligible, the participant will be randomized on Day -1 to receive either AFQ056 or placebo in a 1:1: ratio and at the same time, will also be randomized to a specific couple of sequences saline/cocaine or cocaine/saline for Infusion Session 2 and Infusion Session 3 within each treatment group. The order of the saline and cocaine infusions for each participant for Infusion Sessions 4 and 5 will be the same as the randomized order for Infusion Sessions 2 and 3, respectively.

Participants will receive baseline infusions determined by the randomized sequences of saline and 20 mg of cocaine on Day 1 (Infusion Session 2) and saline and 40 mg of cocaine on Day 2 (Infusion Session 3). The participants will receive either AFQ056 or matching placebo twice a day from Days 3 to 9. The AFQ056 treatment group will be up titrated to 200 mg according to the following dosing schedule: Day 3: 50 mg twice daily; Day 4: 100 mg twice daily and Days 5-9: 200 mg twice daily. On Day 10, participants will be administered only the morning dose of AFQ056 200 mg or placebo. AFQ056 doses must be taken within 30 minutes of meals. On Day 9 and Day 10, approximately 4 hours after the morning dose of AFQ056 200 mg or placebo, participants will receive treatment infusions determined by the randomized sequence of saline and 20 mg of cocaine on Day 9 (Infusion Session 4) and saline and 40 mg of cocaine on Day 10 (Infusion Session 5). The participants will be discharged from the research clinic on Day 12, two days after the last infusion of cocaine (Infusion Session 5) and will have a Follow-up visit between 7 and 14 days after clinic discharge. A safety follow-up call will be conducted 30 days following the last administration of study treatment on Day 40.

ELIGIBILITY:
Key Inclusion Criteria:

* Non-treatment seeking participants who meet DSM-V criteria for cocaine use disorder as assessed using the Mini International Neuropsychiatric Interview (MINI) neuropsychiatric interview (version 7.0).
* Be between 18 and 55 years of age, inclusive
* Have a body mass index (BMI) within a range of 18.0 to 34.0 kg/m2 and a minimum weight of at least 50.0 kg at screening.
* Have experience using cocaine by the smoked or IV route at least 6 times in the past 12 months prior to clinic intake (Day -3) and at least one use within the past 30 days.
* Provide a urine sample positive for cocaine at least once during screening (Days -28 to -4).

Key Exclusion Criteria:

* Have a current or past history of seizure disorder, including alcohol- or stimulant-related seizure, febrile seizure, or significant family history of idiopathic seizure disorder.
* Have any previous medically adverse reaction to cocaine, including loss of consciousness, chest pain, paranoid reaction or seizure.
* Have clinically significant findings in the opinion of an investigator based on the MINI (version 7.0) neuropsychiatric interview.
* Be pregnant or lactating.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception from at least 30 days prior to the first administration of study treatment (Day -2), while taking study treatment, and for at least 30 days after the last dose of the study treatment.
* Have a systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg and heart rate > 100 beats per minute at screening or clinic intake (Day -3).
* Have a history of liver or renal disease or current elevation of aspartate aminotransferase (AST), alanine aminotransferase (ALT) or creatinine, 1.5 × the upper limit of normal at screening or intake (Day -3).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-21 (Estimated); Primary Completion 2022-01-03 (Estimated); Study Completion 2022-01-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events | up to 26 days post-drug administration with a 30-day safety follow-up call
  The distribution of adverse events (AEs) will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.

SECONDARY OUTCOMES:
Observed maximum plasma concentration (Cmax) for cocaine and benzoylecgonine (BE) | Day 2, Day 10
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Area Under the plasma concentration-time Curve from the time 0 to the last observed quantifiable concentration (AUC(0-t)) for cocaine and benzoylecgonine (BE) | Day 2, Day 10
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC(0-t) will be listed and summarized using descriptive statistics.
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) for cocaine and benzoylecgonine (BE) | Day 2, Day 10
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC(0-inf) will be listed and summarized using descriptive statistics.
Time of maximum observed drug concentration occurrence (Tmax) for cocaine and benzoylecgonine (BE) | Day 2, Day 10
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
Terminal rate constant (λz) for cocaine and benzoylecgonine (BE) | Day 2, Day 10
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. λz will be listed and summarized using descriptive statistics.
Terminal elimination half-life (T^1/2) for cocaine and benzoylecgonine (BE) | Day 2, Day 10
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. The half-live will be listed and summarized using descriptive statistics.
Total systemic clearance for intravenous administration (CL) for cocaine and benzoylecgonine (BE) | Day 2, Day 10
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. CL will be listed and summarized using descriptive statistics.
Observed maximum plasma concentration (Cmax) for AFQ056 | Day 10
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Area Under the plasma concentration-time Curve from the time 0 to the last observed quantifiable concentration (AUC(0-t)) for AFQ056 | Day 10
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC(0-t) will be listed and summarized using descriptive statistics.
Area Under the plasma concentration-time Curve From 0 To 12 Hours (AUC0-12) for AFQ056 | Day 10
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC0-12 will be listed and summarized using descriptive statistics.
Time of maximum observed drug concentration occurrence (Tmax) for AFQ056 | Day 10
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
Trough plasma concentration (Ctrough) for AFQ056 | Day 10
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Ctrough will be listed and summarized using descriptive statistics.
Terminal elimination half-life (T^1/2) for AFQ056 | Day 10
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. The half-live will be listed and summarized using descriptive statistics.
Terminal rate constant (λz) for AFQ056 | Day 10
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. λz will be listed and summarized using descriptive statistics.
Apparent clearance of the drug from plasma after oral administration (CL/F) for AFQ056 | Day 10
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. CL/F will be listed and summarized using descriptive statistics.
Visual Analog Scales (VAS) | up through day 10
  The VAS is a self-administered assessment evaluating the subjective effects of cocaine. Participants will use an electronic patient reported outcomes (ePRO) system to answer VAS.
Brief Substance Craving Scale (BSCS) | up through Day 10
  The BSCS is a self-administered assessment that asks the participant to rate his or her craving for cocaine. the BSCS used for this study is a modification of the State of Feelings and Cravings Questionnaire. Participants will use an electronic patient reported outcomes (ePRO) system to answer BSCS.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No